CLINICAL TRIAL: NCT00984477
Title: A Phase I, Exploratory Study to Assess the Pharmacokinetics of Single Oral Doses and a Single Intravenous Radiolabelled Microtracer Dose of AZD5122 in Healthy Male Subjects
Brief Title: Study to Investigate the Activity of AZD5122 When Given as a Single Dose to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2650C00006
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Healthy volunteer; healthy subjects; AZD5122; single oral dose; phase 1; Healthy volunteer phase 1 study
MeSH Terms: interventions — AZD5122

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AZD5122 oral suspension (part A and B)
  Interventions: Drug: AZD5122
- 2 (Placebo Comparator): Placebo oral suspension (part A)
  Interventions: Drug: Placebo
- 3 (Experimental): AZD5122 oral and IV infusion (part B)
  Interventions: Drug: AZD5122

INTERVENTIONS:
Drug: AZD5122 — A single dose of oral suspension
  Arms: 1; 3
Drug: Placebo — A single dose of oral suspension
  Arms: 2
Drug: AZD5122 — A single intravenous infusion
  Arms: 3

SUMMARY:
The purpose of the study is to determine how quickly AZD5122 is absorbed into and cleared by the body when given to healthy, non smoking males at different dose levels. This is a 2 part study, in Part B a single group of subjects will be given both an oral dose and intravenous microdose of AZD5122 at a specialist unit. For part B there is no placebo treatment given.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent.
* Normal physical examination, laboratory values, blood pressure and pulse
* Healthy male caucasian subjects

Exclusion Criteria:

* Subjects must not have any history of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with how drugs are absorbed, used or eliminated by the body.
* Subjects must not have abnormal blood or urine tests for hsCRP, circulating neutrophils, haematocrit, haemoglobin or renal function
* Subjects must not have crystals or more than a trace of blood in their urine

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD5122 in blood | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose.

SECONDARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD5122 in urine | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose.
Measurement of the effect of AZD5122 on circulating neutrophils | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose.
Pharmacodynamic profile: assessment of various pharmacodynamic measures | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 48 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sparrow, BSc, BMedSci, BM,BS, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Queens Medical Centre, Nottingham NG7 2UH
Locations (1):
- Research Site, Nottinghamshire, United Kingdom